CLINICAL TRIAL: NCT01588639
Title: A Prospective Multi-centre, Non-randomized, Open-label, Non-interventional Study to Evaluate the Safety, Efficacy and Injection Compliance of Scilin N, Scilin R or Scilin M30 in Chinese Type 2 Diabetes Mellitus (T2DM)
Brief Title: To Evaluate Clinical Outcome and Injection Compliance of Scilin
Acronym: SEAS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16372; SL1210CN (Other: company internal)
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Recombinant human insulin; T2DM; Safety; Efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Insulin (Scilin N, BAY81-9924); Drug: Insulin (Scilin R _BAY81-9924; Drug: Insulin(Scilin M30_BAY81-9924)

INTERVENTIONS:
Drug: Insulin (Scilin N, BAY81-9924) — Subjects are treated with recombinant human insulin-SciLin N, SciLin R and SciLin M30 (alone or in combination) in routine clinical practice.
Drug: Insulin (Scilin R _BAY81-9924 — Subjects are treated with recombinant human insulin-SciLin N, SciLin R and SciLin M30 (alone or in combination) in routine clinical practice
Drug: Insulin(Scilin M30_BAY81-9924) — Subjects are treated with recombinant human insulin-SciLin N, SciLin R and SciLin M30 (alone or in combination) in routine clinical practice

SUMMARY:
This is a prospective, multi-center, open-label, non-interventional, 12-week study in people with type 2 diabetes mellitus who are treated with recombinant human insulin-SciLin N, SciLin R and SciLin M30 (alone or in combination) in routine clinical practice. The term study insulins will be used in this protocol for these drugs and combinations.

ELIGIBILITY:
Inclusion Criteria:

* Based on physicians' clinical judgement, subjects who are treated with SciLin N, SciLin R and SciLin M30 ( alone or in combination) will be eligible to be included in this clinical study.

Exclusion Criteria:

Subjects with one of the conditions listed below will be excluded:

Women who are pregnant, breast feeding or have the intention of becoming pregnant within the next 6 months Subjects who have to be treated with other insulins simultaneously Subjects who are participating in other diabetes clinical studies at the same time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 2683 (Actual)
Dates: Start 2012-08; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Occurrence rate of serious adverse drug reactions including severe hypoglycaemic events | up to 12 week

SECONDARY OUTCOMES:
Occurrence rate of hypoglycemic events | up to 12 weeks
Change in HbA1c | Baseline and week 12
Change in FPG (Fasting Plasma Glucose) | Baseline and week 12
Change in PPG (Postprandial Glucose) | Baseline and week 12
The ratio of compliance injection (following physician's advice) | up to 12 weeks
Number and ratio of missed injections | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, China